CLINICAL TRIAL: NCT00967447
Title: Incidence of Symptomatic Venous Thromboembolic Events and Major Bleeding Events After Dabigatran Etexilate in Patients Subject to Subject to Elective Total Hip or Knee Replacement Surgery.
Brief Title: Study to Evaluate the Safety and Efficacy of Pradaxar for the Prevention of Venous Thromboembolism in the Mexican Population Undergoing Elective Total Hip or Knee Replacement Surgery
Status: Terminated | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1160.103
Record Dates: First submitted 2009-08-13; First posted 2009-08-27 (Estimated); Results first posted 2012-04-05 (Estimated); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: Thromboembolism; Arthroplasty, Replacement, Hip
MeSH Terms: conditions — Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Open, prospective, uncontrolled, observational cohort study.

ELIGIBILITY:
Inclusion criteria:

* patients age 18 years or above undergoing elective total hip or knee replacement surgery
* Written informed consent obtained for data collection and source data verification.

Exclusion criteria:

According to the approved label the following patients should not be treated with Pradaxar® 220mg q.d.:

* age of > 75 years
* renal impairment (creatinine clearance <50ml/min)
* patients on concomitant therapy with amiodarone or verapamil.
* elevated liver enzymes >2 upper limit of normal (ULN) and / or hepatic impairment or liver disease expected to have any impact on survival
* anaesthesia with post-operative indwelling epidural catheters
* hypersensitivity to dabigatran etexilate or to any of the excipients
* active clinically significant bleeding
* organic lesion at risk of bleeding
* spontaneous or pharmacological impairment of haemostasis except for the above-included patients groups
* concomitant treatment with quinidine

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinics
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2009-02-01 (Actual); Primary Completion 2010-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (28):
- Mexico (28):
  - Boehringer Ingelheim Investigational Site 10, Distrito Federal
  - Boehringer Ingelheim Investigational Site 11, Distrito Federal
  - Boehringer Ingelheim Investigational Site 12, Distrito Federal
  - Boehringer Ingelheim Investigational Site 13, Distrito Federal
  - Boehringer Ingelheim Investigational Site 14, Distrito Federal
  - Boehringer Ingelheim Investigational Site 15, Distrito Federal
  - Boehringer Ingelheim Investigational Site 16, Distrito Federal
  - Boehringer Ingelheim Investigational Site 17, Distrito Federal
  - Boehringer Ingelheim Investigational Site 18, Distrito Federal
  - Boehringer Ingelheim Investigational Site 19, Distrito Federal
  - Boehringer Ingelheim Investigational Site 1, Distrito Federal
  - Boehringer Ingelheim Investigational Site 20, Distrito Federal
  - Boehringer Ingelheim Investigational Site 2, Distrito Federal
  - Boehringer Ingelheim Investigational Site 3, Distrito Federal
  - Boehringer Ingelheim Investigational Site 4, Distrito Federal
  - Boehringer Ingelheim Investigational Site 5, Distrito Federal
  - Boehringer Ingelheim Investigational Site 6, Distrito Federal
  - Boehringer Ingelheim Investigational Site 7, Distrito Federal
  - Boehringer Ingelheim Investigational Site 8, Distrito Federal
  - Boehringer Ingelheim Investigational Site 9, Distrito Federal
  - Boehringer Ingelheim Investigational Site 21, Guadalajara
  - Boehringer Ingelheim Investigational Site 22, Guadalajara
  - Boehringer Ingelheim Investigational Site 23, Guadalajara
  - Boehringer Ingelheim Investigational Site 24, Guadalajara
  - Boehringer Ingelheim Investigational Site 25, Guadalajara
  - Boehringer Ingelheim Investigational Site 28, Monterrey
  - Boehringer Ingelheim Investigational Site 26, Puebla City
  - Boehringer Ingelheim Investigational Site 27, Puebla City

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only two patients were included into the study. The sponsor decided to finish it due to a delay of recruitment period.
Groups:
- Dabigatran Exilate 220 Once Daily (OD): 10 days for Knee Replacement or 28-35 Hip Replacement
Period: Overall Study
Arm/Group | Dabigatran Exilate 220 Once Daily (OD)
Started | 2 (there are no collected data in CRF)
Completed | 2 (there are no collected data in CRF)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Dabigatran Exilate 220 Once Daily (OD)
Number analyzed (Participants) | 0
Age, Continuous [unit: years]
Sex: Female, Male

OUTCOME MEASURES:

1. Primary Outcome: Venous Thromboembolic Events
Time Frame: 6 Months
Population: The trial was stopped due poor enrollment
Arm/Group | Dabigatran Exilate 220 Once Daily (OD)
Number analyzed (Participants) | 0

2. Secondary Outcome: Major Bleeding Events (MBE)
Time Frame: From 12 To 37 Days
Population: The trial was stopped due poor enrollment
Arm/Group | Dabigatran Exilate 220 Once Daily (OD)
Number analyzed (Participants) | 0

3. Secondary Outcome: Major Extra Surgical Site Bleedings
Time Frame: From 12 To 37 Days
Population: The trial was stopped due poor enrollment
Arm/Group | Dabigatran Exilate 220 Once Daily (OD)
Number analyzed (Participants) | 0

4. Secondary Outcome: Volume of Wound Drainage
Time Frame: From 12 To 37 Days
Population: The trial was stopped due poor enrollment
Arm/Group | Dabigatran Exilate 220 Once Daily (OD)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Dabigatran Exilate 220 Once Daily (OD)
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the results of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract